CLINICAL TRIAL: NCT00099424
Title: EXercise TRAining in Sarcoidosis (EXTRAS Study): A Prospective, Randomized, Controlled, Crossover Trial
Brief Title: Exercise Training in Sarcoidosis (EXTRAS Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: ML2563
Record Dates: First submitted 2004-12-13; First posted 2004-12-14 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Sarcoidosis
Keywords: exercise training; resistance training; endurance training; Boeck's Sarcoid; Besnier-Boeck Disease
MeSH Terms: conditions — Sarcoidosis

INTERVENTIONS:
Behavioral: High-intensity exercise training

SUMMARY:
Exercise intolerance and reduced health status have been found in patients with sarcoidosis and has been related to skeletal muscle weakness. The present researchers reason that skeletal muscle weakness is, at least in part, related to physical inactivity and therefore partially reversible following a structured exercise training program. Nevertheless, the effects of exercise training have never been studied in patients with sarcoidosis. Therefore, the present study is undertaken to explore the effects of exercise training in patients with sarcoidosis. A priori, the following hypotheses are formulated:

* A 12-week exercise training program improves health status, quality of life and exercise capacity in patients with sarcoidosis as compared to sarcoidosis patients without exercise intervention.
* A 12-week exercise training program improves skeletal muscle function and reduces complaints of anxiety and depression in patients with sarcoidosis as compared to sarcoidosis patients without exercise intervention.
* A 12-week exercise training program reduces circulating levels of inflammatory markers in patients with sarcoidosis as compared to sarcoidosis patients without exercise intervention.

DETAILED DESCRIPTION:
The EXTRAS study is a prospective, randomized, controlled, 24-week crossover clinical trial in which the participants are randomly assigned to receive 12 weeks of dynamic resistance and whole-body endurance exercises followed by 12 weeks without intervention or vice versa. Consenting participants will be assessed at baseline (before randomization, week 0) and at weeks 12 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Main diagnosis: previously diagnosed sarcoidosis according to the latest ATS/ERS/WASOG statement on sarcoidosis (AJRCCM 1999)

Exclusion Criteria:

* A history of neurosarcoidosis
* Undergoing structured exercise training at the time of enrollment or in the preceding 6 months
* Current participation in a pharmacological study
* Cardiovascular abnormalities on the ECG during baseline peak exercise test
* A 'normal' baseline peak oxygen uptake (≥90% of the predicted values) in combination with a 'normal' quadriceps peak torque or distance walked in 6 minutes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-02; Study Completion 2005-08

PRIMARY OUTCOMES:
Health status: Medical Outcomes Study 36-Item Short-Form Health Survey
Disease-specific quality of life: Sarcoidosis Health Questionnaire
Peak exercise capacity: a symptom-limited peak exercise test on a cycle ergometer
Functional exercise capacity (I): a symptom-limited endurance cycling test at 70% of the achieved peak external load
Functional exercise capacity (II): the distance walked in 6 minutes

SECONDARY OUTCOMES:
Pulmonary function: forced vital capacity and transfer factor for carbon monoxide
Muscle function: isometric quadriceps femoris muscle peak torque
Systemic inflammation: circulating levels of IL-2, sIL-2r, IL-6, IL-8, TNF-alpha, sTNFR-p55, sTNFR-p75
Anxiety and depression: Hospital Anxiety and Depression Scale
Health-related quality of life (I): Chronic Respiratory Disease Questionnaire
Health-related quality of life (II): St. George's Respiratory Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Martijn A. Spruit, PhD, Principal Investigator — KU Leuven; Marc Decramer, PhD MD, Study Director — University Hospital, Gasthuisberg; Michiel J. Thomeer, MD, Study Chair — University Hospital, Gasthuisberg
Locations (1):
- University Hospital Leuven, Leuven, Vlaams-Brabant, Belgium